CLINICAL TRIAL: NCT07051902
Title: Analyzing the Microbiome and Environmental Exposures of Patients Suffering From Atopic Diseases in Mali
Brief Title: Microbiome and Atopy in Mali
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Microbiome in Mali
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Atopic Disease
Keywords: asthma; atopic dermatitis; allergies
MeSH Terms: conditions — Asthma; Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin swabs, nasal swabs, sputum, whole blood, stool, urine, skin tape strip
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with atopic disease (asthma or atopic dermatitis)
- Age/sex-matched healthy volunteers.

SUMMARY:
This study is about allergic diseases in people living in Mali. Allergic diseases can cause health problems like asthma or skin rashes. In this study, we will look for clues about things that may affect whether people get allergic diseases. We will look at things on or in the body, like germs, and things in the environment, like pollution. To do this, we will collect different types of biological samples, health information, and environmental information from people with allergic diseases and people without allergic diseases. We will compare what we find in each group to look for differences that might be related to allergic disease.

DETAILED DESCRIPTION:
This is a case-control study where participants from Bamako in Mali will be screened to identify patients with atopic disease (asthma and atopic dermatitis). Age and sex-matched healthy controls will be selected at a 1:1 ratio. All study participants (including healthy controls) will undergo a clinical evaluation and provide skin swabs, nasal swabs, induced sputum (if successful), blood samples, drinking water samples, stool samples, as well as complete an interviewer-administered questionnaire on environmental exposures. All participants (including healthy controls) will also undergo pulmonary function testing (spirometry and/or oscillometry) and undergo testing of transepidermal electrical impedance (using a Nevisense machine). Samples will be used to evaluate the microbiome diversity in participants with allergy-related diseases (ARDs) compared to healthy controls. Environmental surveys will assess the association between atopy and exposures that are primarily outdoor versus indoor exposures. Temporal and spatial variation in these pollutants will be assessed. Air samples taken from the community and participant home drinking water samples (when available) will be used to assess the presence and variability of pollutants in the environment.

ELIGIBILITY:
Inclusion Criteria (Study Group):

* Aged ≥3 years.
* Able to provide informed consent (for ages ≥18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 years).
* Positive Screening questionnaire for asthma or eczema.
* Diagnosed with atopic dermatitis or asthma via physician diagnosis and criteria as follows:
* Clinical diagnosis of atopic disease, as defined by Hanifin and Rajka criteria, that has been present for ≥3 months before the screening visit.

Inclusion Criteria (Healthy Volunteers):

* Aged ≥3 years.
* Able to provide informed consent (for ages ≥18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 years).
* Negative Screening questionnaire for asthma and eczema.
* In good general health as evidenced by medical history and not diagnosed with atopic dermatitis or asthma via physician diagnosis.
* Failure to meet Hanifin and Rajka criteria and <3 on GINA guidelines for asthma diagnosis.
* No self-reported history of food allergy.

Exclusion Criteria:

* Use of antibiotics in the 3 months prior to screening.
* Current pregnancy or lactation (determined by self-report).
* Treatment with an investigational drug within 12 months prior to screening.
* Current smoker or tobacco use within 4 months prior to screening.
* Current skin infections other than atopic dermatitis (e.g., scabies).
* Active diarrhea as defined by three or more loose stools per day (Bristol stool scale score of 6 or 7).
* Presence of current bacterial, viral, or fungal infection, with the exception of isolated onchomycosis, which is not exclusionary.
* Any other condition or factor that the investigator determines may significantly influence the results of testing.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited from the Bamako area
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Differences in gut microbiome between atopic patients and healthy controls in children and adults. | Within 28 days after the screening visit.
  Shannon diversity index analyzed using t-test with significance level of .05.

SECONDARY OUTCOMES:
Relative abundance of taxa and expression of metabolically functional genes in the skin microbiome. | Within 28 days after the screening visit.
  RNAseq
Relative abundance of taxa and expression of metabolically functional genes in the gut microbiome. | Within 28 days after the screening visit.
  Metagenomic sequencing
Relative abundance of taxa and expression of metabolically functional genes in the nasal microbiome | Within 28 days after the screening visit.
  Metagenomic sequencing
Presence, frequency, and/or proximity to environmental exposures. | Within 28 days after the screening visit.
  Patient survey
Serum concentration of total IgE, specific IgE panels, and eosinophils | Within 28 days after the screening visit.
Concentration of pollutants or pollutant biomarkers in urine and serum | Within 28 days after the screening visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Shobnam, MD, Principal Investigator — LCIM, NIAID, NIH; Ian Myles, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Mali (2):
  - Dermatology Hospital of Bamako, Bamako
  - Pneumology Ward, Point G University Hospital, Bamako